CLINICAL TRIAL: NCT06532552
Title: Comparison of VA (Venetoclax, Azacitidine), VACl (VA, Cladribine), VACh (VA, Chidamide), and Alternating VACl/VACh in Newly Diagnosed Adult Acute Myeloid Leukemia Patients Ineligible for Intensive Therapy or Declining: A Prospective, Multi-center, Randomized, Controlled Phase II Study
Brief Title: Comparison of VA (Venetoclax, Azacitidine), VACl (VA, Cladribine), VACh (VA, Chidamide), and Alternating VACl/VACh in Newly Diagnosed Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Jining Medical University (Other); Qilu Hospital of Shandong University (Other); The Affiliated Hospital of Qingdao University (Other); The First Affiliated Hospital of Anhui Medical University (Other); Tongji Hospital (Other); The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, professor, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZAML06
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia, Adult; Newly Diagnosed
Keywords: Venetoclax; Azacitidine; Cladribine; Chidamide
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VA group (Active Comparator): Azacitidine 75mg/m2 subcutaneous daily for 7 days and Venetoclax orally once daily (100mg d1, 200mg d2, 400mg d3-28). Patients received 2 cycles of VA, the bone marrow aspirate will be done on the 21-28th day in the each cycle. If the result is partial remission (PR)/no response (NR) at the end of the cycle 2, the patients need to withdraw from the trial. If the bone marrow assessment is complete remission (CR)/CR with incomplete hematologic recovery (CRi)/morphologic leukemia-free state (MLFS), the patients will start post-remission therapy. For post-remission therapy, if the patients ineligible for intensive chemotherapy or declines, continue with the same regimen until progression or recurrence of the disease, and the patients need to withdraw from the trial. If the patients fit for intensive chemotherapy, patients will receive chemotherapy with other regimens or transplantation, and the patients need to withdraw from the trial if progression or recurrence of the disease.
  Interventions: Drug: VA
- VACl group (Experimental): Azacitidine 75mg/m2 subcutaneous Daily for 7 days, Venetoclax orally once daily (100 mg d1, 200mg d2, 400mg d3-28) and Cladribine 5mg/m2 intravenous (IV) over approximately 1 to 2 hours, daily on days 1-3. Patients received 2 cycles of VACl treatments, the bone marrow aspirate will be done on the 21-28th day in the each cycle. If the bone marrow assessment is PR/NR at the end of the cycle 2, the patients need to withdraw from the trial. If the bone marrow assessment is CR/CRi/MLFS, the patients will start post-remission therapy. For post-remission therapy, if the patients ineligible for intensive chemotherapy or declines, continue with the same regimen until progression or recurrence of the disease, and the patients need to withdraw from the trial. If the patients fit for intensive chemotherapy, patients will receive consolidation chemotherapy with other regimens or transplantation, and the patients need to withdraw from the trial if progression or recurrence of the disease.
  Interventions: Drug: VACl
- VACh group (Experimental): Azacitidine 75mg/m2 subcutaneous daily for 7 days, Venetoclax orally once daily (100mg d1, 200mg d2, 400mg d3-28) and Chidamide 10mg orally daily for 12 days. Patients received 2 cycles of VACh treatments, the bone marrow aspirate will be done on the 21-28th day in the each cycle. If the bone marrow assessment is PR/NR at the end of the cycle 2, the patients need to withdraw from the trial. If the bone marrow assessment is CR/CRi/MLFS, the patients will start post-remission therapy. For post-remission therapy, if the patients ineligible for intensive chemotherapy or declines, continue with the same regimen until progression or recurrence of the disease, and the patients need to withdraw from the trial. If the patients fit for intensive chemotherapy, patients will receive consolidation chemotherapy with other regimens or transplantation, and the patients need to withdraw from the trial if progression or recurrence of the disease.
  Interventions: Drug: VACh
- VACl Alternating With VACh group (Experimental): Patients received 1 cycle of VACl and 1 cycle of VACh treatment, the bone marrow aspirate will be done on the 21-28th day in the each cycle. If the bone marrow assessment is PR/NR at the end of the cycle 2, the patients need to withdraw from the trial. If the bone marrow assessment is CR/CRi/MLFS, the patients will start post-remission therapy. For post-remission therapy, if the patients ineligible for intensive chemotherapy or declines, continue with the VACl alternating with VACh until progression or recurrence of the disease, and the patients need to withdraw from the trial. If the patients fit for intensive chemotherapy, patients will receive consolidation chemotherapy with other regimens or transplantation, and the patients need to withdraw from the trial if progression or recurrence of the disease.
  Interventions: Drug: VACl Alternating With VACh

INTERVENTIONS:
Drug: VACl — Azacitidine:75mg/m2 Subcutaneous daily for 7 days Venetoclax: orally once daily (100 mg d1, 200mg d2, 400mg d3-28) Cladribine: 5mg/m2 IV over approximately 1 to 2 hours, daily on days 1-3.
  Other Names: Venetoclax+Azacitidine+Cladribine
  Arms: VACl group
Drug: VACh — Azacitidine: 75mg/m2 Subcutaneous daily for 7 days Venetoclax: orally once daily (100mg d1, 200mg d2, 400mg d3-28) Chidamide: 10mg orally daily for 12 days
  Other Names: Venetoclax+Azacitidine+Chidamide
  Arms: VACh group
Drug: VACl Alternating With VACh — VACl:
  Azacitidine:75mg/m2 Subcutaneous daily for 7 days Venetoclax: orally once daily (100 mg d1, 200mg d2, 400mg d3-28) Cladribine: 5mg/m2 IV over approximately 1 to 2 hours, daily on days 1-3.
  VACh:
  Azacitidine: 75mg/m2 Subcutaneous daily for 7 days Venetoclax: orally once daily (100mg d1, 200mg d2, 400mg d3-28) Chidamide: 10mg orally daily for 12 days
  Other Names: Venetoclax+Azacitidine+Cladribine alternating with Venetoclax+Azacitidine+Chidamide
  Arms: VACl Alternating With VACh group
Drug: VA — Azacitidine: 75mg/m2 Subcutaneous (SC) daily for 7 days Venetoclax: orally once daily (100mg d1, 200mg d2, 400mg d3-28).
  Other Names: Venetoclax+Azacitidine
  Arms: VA group

SUMMARY:
This prospective, multi-center, randomized, controlled Phase II study is to compare the therapeutic efficacy and side effect of VACl (Venetoclax,Azacitidine,Cladribine) alternating with VACh (Venetoclax,Azacitidine,Chidamide), VACl, VACh and VA in newly diagnosed adult acute myeloid leukemia (AML) patients ineligible for intensive therapy or declining. Cladribine is a purine analogue widely used in hematologic malignancies. The monocytic leukemia stem cell is selective sensitivity to Cladribine. Chidamide, a newly designed selective histone deacetylase inhibitor, could down regulate myeloid cell leukaemia 1 (MCL1) expression in Venetoclax resistant AML cells. Chidamide or Cladribine have synergistic anti-leukemia effects with VA through their unique mechanisms, which can eradicate leukemia stem cells and prevent the occurrence of drug resistance.

DETAILED DESCRIPTION:
AML is a clonal myelopoietic stem cell disorder characterized by the accumulation of neoplastic cells in the bone marrow and in the peripheral circulation. The median age of AML patients is 68 years. Although intensive chemotherapy and allogeneic stem cell transplant (allo-HSCT) are standard approaches for newly diagnosed patients, they are associated with higher rates of treatment related complications and inferior outcomes in older patients. Venetoclax, a newly orally available and selective B cell lymphoma-2 (BCL2) inhibitor, Venetoclax in combination with hypomethylation agents or cytarabine has been approved by the Food and Drug Administration (FDA) for the treatment of patients with newly diagnosed AML unfit for intensive chemotherapy. However, the emergence of resistance to Venetoclax based combinations has become an important clinical dilemma. Resistance to Venetoclax can be acquired through the up regulation of anti-apoptotic proteins, such as myeloid cell leukaemia 1 (MCL1). Chidamide, a newly designed selective histone deacetylase inhibitor, Chidamide could down Bregulate MCL1 expression in Venetoclax resistant AML cells. Our experience showed that the Chidamide+VA could improve the condition of R/R AML patients who are resistant to VA. Cladribine is a purine analogue widely used in hematologic malignancies. It was demonstrated that addition of Cladribine to the VA regimen increases eradication of primary AML containing monocytic leukemia stem cell activity in both in vitro and in vivo preclinical models. Chidamide or Cladribine have synergistic anti-leukemia effects with VA through their unique mechanisms, which can eradicate leukemia stem cells and prevent the occurrence of drug resistance, thereby increasing response rate, prolonging patient survival, reducing recurrence, and improving prognosis without increasing treatment-related complications. Therefore, this prospective, multi-center, randomized, controlled Phase II study is to compare the therapeutic efficacy and side effect of VACl (Venetoclax,Azacitidine,Cladribine) alternating with VACh (Venetoclax,Azacitidine,Chidamide), VACl, VACh and VA in newly diagnosed adult AML patients ineligible for intensive therapy or declining.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for study participation if he/she meets the following criteria within 21 days prior to randomization.

1. Subject must have confirmation of previously untreated AML by World Health Organization (WHO) criteria, and be ineligible for treatment with a standard cytarabine and anthracycline induction regimen due age or comorbidities. Prior therapy with hydroxyurea or a total dose of cytarabine no more than 0.5g (for emergency use for stabilization) is allowed.
2. Subject must be≥18 years of age with at least one of the following conditions:

   A)≥60 years of age; B) Patients aged < 60 years who are unsuitable for standard induction therapy（Any other comorbidity that the physician judges to be incompatible with conventional intensive chemotherapy); C) The patient refused the conventional intensive chemotherapy.
3. Adequate organ function as defined below:

   A)liver function (bilirubin≤2mg/dL, aspartate transaminase (AST) and/or alanine transaminase (ALT)≤3 x ULN).

   Unless liver enzyme abnormalities are determined by the treating MD and PI to be due to leukemic infiltration.

   B)kidney function (creatinine≤1.5xULN ).
4. ECOG performance status of ≤ 2.
5. A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.
6. Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient or his legally authorized representative is required prior to their enrollment on the protocol.
7. Patient must have a projected life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Subject has a history of other malignancies prior to study entry, with the exception of:

   A) Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast; B) Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; C) Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
2. Subject has acute promyelocytic leukemia, subject has history of myeloproliferative neoplasm [MPN] including myelofibrosis, essential thrombocythemia, polycythemia vera, CML with or without BCR-ABL1 translocation, BCR/ABL positive AML.
3. Patient has known active central nervous syster (CNS) involvement with AML.
4. Subject has a white blood cell count> 25×10^9/L. (Hydroxyurea is permitted to meet this criterion.)
5. Prior therapy with venetoclax, Cladribine, hypomethylating agents (HMAs), Chidamide or Chimeric Antigen Receptor T cell therapy, experimental therapies for MDS or AML.
6. Subject has a malabsorption syndrome or other condition that precludes enteral route of administration.
7. Subject is known to be positive for human immunodeficiency virus (HIV) (HIV testing is not required.)
8. Subject has received strong and/or moderate CYP3A inducers within 7 days prior to the initiation of study treatment.
9. Subject has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Starfruit within 3 days prior to the initiation of study treatment.
10. Subject has a cardiovascular disability status of New York Heart Association Class≥2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or anginal pain.
11. Subject has chronic respiratory disease that requires continuous oxygen, or significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, or any other medical condition that in the opinion of the investigator would adversely affect his/her participating in this study.
12. Subject exhibits evidence of other clinically significant uncontrolled systemic infection requiring therapy (viral, bacterial or fungal).
13. Subject is known to be positive for hepatitis B or C infection with the exception of those with an undetectable viral load within 3 months (Hepatitis B or C testing is not required). Subjects with serologic evidence of prior vaccination to HBV [i.e., HBs Ag-, and anti-HBs+-] may participate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 1 year
  It is defined as the number of days from the date of randomization to the date of earliest evidence of relapse, subsequent treatment other than stem cell transplant while in composite complete remission (CR+CRi), or death. If the specified event (relapse, start of subsequent treatment, or death) does not occur, subjects will be censored at the date of last disease assessment.
Cumulative incidence of relapse (CIR) | 1 year
  Time from CR to disease recurrence or progression

SECONDARY OUTCOMES:
Composite complete response (CRc) | At the end of Cycle 1 (each cycle is 21-28 days)
  CRc rate was defifined as patients achieving a CR or CRi
Overall Survival (OS) | 1 year
  Time from date of treatment start until date of death due to any cause
Adverse reactions in hematology | At the end of Cycle 1 (each cycle is 21-28 days)
  Record of adverse events in hematological system during and after VA,VACl,VACh,VACl alternating with VACh regimen induction (agranulocytosis days, platelet（PLT）/red blood cell (RBC) transfusion units)
Nonhematological adverse reactions | At the end of Cycle 1 (each cycle is 21-28 days)
  Record of adverse events in other organs or systmes during and after VA,VACl,VACh,VACl alternating with VACh regimen induction (infection and organ injury)

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Li Xue, M.D., Principal Investigator — The First Affliated Hospital of Soochow University
Locations (1):
- The First Affliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No